CLINICAL TRIAL: NCT05534126
Title: Enhancing Cognitive Processing Therapy for Posttraumatic Stress Disorder Via Stellate Ganglion Block Treatment: A Pilot Trial
Acronym: SGB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Philip Held, Research Director, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22011306
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Posttraumatic Stress Disorder; Chronic Pain
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate Ganglion Block (Active Comparator)
  Interventions: Procedure: Stellate Ganglion Block Treatment
- Placebo (Placebo Comparator)
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Stellate Ganglion Block Treatment — Stellate ganglion block procedure is a treatment that involves injection of local anesthetic around the stellate ganglion (located at the base of the neck) to block its transmission of pain signals.
  Arms: Stellate Ganglion Block
Procedure: Placebo — Sham
  Arms: Placebo

SUMMARY:
Cognitive Processing Therapy (CPT) is an effective first-line, evidence-based treatment for posttraumatic stress disorder (PTSD). Despite its well-demonstrated effectiveness, research has shown that approximately two-thirds of individuals continue to meet the diagnostic criteria for PTSD even after successful treatment completion. Stellate Ganglion Block (SGB) treatment, involving a local anesthesia injection to the stellate ganglion (around the lower base of the neck), has been shown to block its pain signal transmissions. Prior case studies and reviews have provided evidence for reducing PTSD symptoms with SGB treatment. However, studies to date have only examined SGB as a standalone intervention. The utility of combining CPT with concurrent SGB treatment remains unknown, although it is plausible that the combination of the two treatments can improve the effectiveness of CPT alone. The present study aims to test this hypothesis by comparing either a combined 1-week massed CPT + SGB treatment and 1-week massed CPT + placebo treatment (saline injection) using a randomized controlled trial design.

ELIGIBILITY:
Inclusion Criteria:

1. Are 18 years or older
2. Are fluent in English
3. Reside in Illinois
4. Have safe transportation means other than driving themselves to Rush University Medical Center for two separate procedures (e.g., Uber, family or friend to drive them to study visits, etc.)
5. Have experienced a Criterion A traumatic event during their lifetime
6. Have a PTSD diagnosis verified via the Clinician Administered PTSD Scale for DSM-5
7. Have not previously received stellate ganglion blocks
8. Are willing and able to participate in daily Cognitive Processing Therapy over the course of one week
9. Are willing and able to complete self-report measures and clinician-rated assessments at multiple time points over the course of the study

Exclusion Criteria:

1. The traumatic event occurred in the past month
2. They are currently suicidal or homicidal (i.e., plan and intent)
3. They have unmanaged psychosis or mania
4. They have not been on a stable dose of psychotropic medication for at least one month by the time of the baseline assessment or are planning to change their medications within 3 months of starting their participation in the study
5. They have completed an evidence-based cognitive behavioral PTSD treatment (e.g., Cognitive Processing Therapy or Prolonged Exposure) in the past 12 months or are currently receiving an evidence-based PTSD treatment
6. They have an intellectual disability or significant cognitive impairment that would prevent them from engaging in CPT, as assessed via the Mini-Mental State Exam-Second Edition (MMSE-2)
7. They are currently on any blood-thinning medications or have a coagulopathy
8. They have any of the following conditions: a recent myocardial infarction, glaucoma, a pre-existing contralateral nerve palsy, severe emphysema or a cardiac conduction blockade.
9. They are allergic to any of the medications injected (i.e., ropivacaine, lidocaine, propofol, medications)
10. They have an active infection
11. They have a serious or unstable medical illness or instability for which hospitalization may be likely within the next year
12. They have a visual or auditory impairment that would prevent them from fully participating in study activities
13. They are involved with current legal actions related to the traumatic event that is anticipated to be targeted during treatment
14. Subjects who, at the time of consent, appear to have extenuating life circumstances (e.g., unstable housing, no internet access, etc.) which, in the judgement of the Principal Investigator, could affect the ability to deliver the intervention with fidelity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale for DSM-5 | Through study completion, on average of 3 months
  Clinician Administered Assessment of PTSD
PTSD Checklist for DSM-5 Criteria | Through study completion, on average of 3 months
  Self-report measure for PTSD

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No